CLINICAL TRIAL: NCT02335138
Title: Project Nexus: Providing Online Counseling for Home-Based HIV Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Miami (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Robert Stephenson, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00072655
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Couples
Keywords: HIV; MSM; Couples; Home Testing; Sexual Agreements
MeSH Terms: interventions — Counseling; chitinase C

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Placebo Comparator): Each participant will receive an at-home test kit and will be asked to test and return results to investigator.
  Interventions: Behavioral: at-home test kit
- Intervention Arm (Active Comparator): Each participant will receive an at-home test kit and will be asked to take the test in conjunction with an online CHTC session.
  Interventions: Behavioral: Couples HIV Testing and Counseling (CHTC, CVCT)

INTERVENTIONS:
Behavioral: Couples HIV Testing and Counseling (CHTC, CVCT) — Male couples randomized to the experimental group (Couples HIV Testing and Counseling, CHTC/CVCT) will receive HIV counseling and testing as a couple via an online, HIPPA-compliant videoconferencing service. The dyad-centered session will last less than one hour and focus on couples agreement, prevention strategies, and/or linkage to HIV care, depending on each couple's test results. Participants will complete follow-up surveys at 3 and 6 months post-testing.
  Other Names: CHTC, CVCT
  Arms: Intervention Arm
Behavioral: at-home test kit — Male couples in the control group will receive test kits, but will not receive any testing intervention. Once individual results are reported,participants will be contacted via phone by study staff with options for referrals to services for the reactive partner(s). Participants will complete follow-up surveys at 3 and 6 months post-testing.
  Arms: Control Arm

SUMMARY:
The proposed research aims to address the question: Compared to the current standard of care for home-based HIV tests, in which persons conduct and interpret HIV tests without counseling, does the addition of video conferencing with a remote counselor increase health-enhancing, protective behaviors among male-male couples and facilitate linkage to care for those who test positive?

DETAILED DESCRIPTION:
The investigators propose to address four specific aims through a randomized controlled trial (RCT) to take place over a four-year period. The investigators plan to enroll and maintain a cohort of 350 men who have sex with men (MSM) couples: 175 self-reported concordant HIV-negative and 175 self-reported HIV-discordant couples. Within this sample, the proposed study will examine the impact of home-testing with video-based Couples HIV Testing and Counseling (CHTC) (intervention) versus home-testing alone (control) on changes in: sexual risk-taking (e.g., UAI), formation and adherence to explicit agreements about sex, relationship functioning for the management of HIV risk, and linkage to care for newly diagnosed HIV positives among MSM couples who live throughout the US. To assess these specific changes, couples will complete online surveys at 3 time points (baseline, 3 months and 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Male sex at birth
* Male gender
* 18 or older
* In a relationship with a male sexual partner of duration six months or longer
* Negative or unknown HIV status and not having tested in the last 6 months, with a partner meeting the same criteria OR in a sero-discordant with the negative/unknown partner reporting not having tested in the past 6 months
* No recent (past year) severe intimate partner violence (IPV) reported within the couple. IPV will be determined by responses to the below questions, in addition to parallel questions addressing perpetration of the specified acts:

  1. Excluding consensual acts such as mutually agreed upon BDSM, in the past year, how many times has [your partner] punched, hit, or slapped you?
  2. Excluding consensual acts such as mutually agreed upon BDSM, in the past year, how many times has [your partner] kicked you?
  3. Excluding consensual acts such as mutually agreed upon BDSM, in the past year, how many times has [your partner] used force or threats of force to make you do something sexual that you didn't want to do?
  4. Excluding consensual acts such as mutually agreed upon BDSM, in the past year, how many times has [your partner] raped you? [Follow up question: Do you feel safe in your relationship?]
* Willingness to have HIV test kits delivered to a home address they provide
* Willingness to be tested for HIV with one's male sexual partner
* Willingness to be randomized to either study arm
* Willingness and ability to participate in video-based counseling (must have a computer or tablet with video and audio capabilities, Internet access)

Exclusion Criteria:

* Sex at birth other than male
* Gender other than male
* Either partner aged 17 or younger
* Does not have a main male sex partner or has a main male sex partner of relationship duration less than 6 months
* Both partners within the couple report known, positive HIV status OR one or both partners reports having tested negative for HIV within 6 months
* Either partner reports experiencing or perpetrating intimate partner violence within the couple within the past year
* Either partner expresses unwillingness to have HIV test kits delivered to a home address
* Either partner expresses unwillingness to test for HIV together with his male sexual partner
* Either partner expresses unwillingness to be randomized
* Unwillingness or inability to participate in video-based counseling

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2016-04; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Process and use of communal coping - Outcome Efficacy to Reduce HIV Threat | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure process and use of communal coping or how couples work together and make decisions together to reduce the health threat. We created three subscales to capture the full range of outcome efficacy related to these three processes of communal coping. For the first subscale, Joint Effort, we used the stem, "My partner and I believe that 'working together' versus on our own is an effective strategy;" for the second subscale, Communication, we used the stem, "Communicating with my partner is an effective strategy for;" and for the third subscale, Planning and Decision-making, we used the stem, "My partner and I making decisions together rather than separately is an effective strategy." The items for each of the three subscales were the same as the items used for the Preference for Sexual Health Outcomes scale.
Process and use of communal coping - Couple Efficacy to Reduce HIV Threat | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure process and use of communal coping or how couples work together and make decisions together to reduce the health threat. Couple efficacy is defined as a couple's confidence that together they can engage in communal coping efforts. We developed three subscales in parallel to Outcome Efficacy to Reduce HIV Threat Scale: Joint Effort, Communication, and Planning and Decision-making.
Process and use of communal coping - Communal Coping to Reduce HIV Threat | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure process and use of communal coping or how couples work together and make decisions together to reduce the health threat. Scale: We developed three subscales in parallel to the Outcome Efficacy Scale and the Couple Efficacy Scale: Joint Effort, Communication, and Planning and Decision-making. All three subscales used the same six items from these other scales to capture the managing of reducing the health threat of HIV, but the stems were different.
Changes in Sexual Agreements | 6 months
  We measure changes in sexual agreements using questions from previous studies of MSM couples' sexual agreements. Participants will be asked which of the following best describes their current sexual agreement with their main partner: "both of us cannot have sex with outside partners," "we can have sex with outside partners, without any conditions or restrictions," "we can have sex with outside partners, but with conditions or restrictions," and "we do not have an agreement." Additional items about agreements will further assess whether couples permitted (or did not permit) that certain sexual behaviors, namely UAI and oral sex, could occur with outside partners. In follow-up surveys, participants will be asked whether their agreement changed, and if so, to re-categorize their agreement type.
Changes in Sexual Behavior | 6 months
  We measure changes in sexual behavior using behavioral measures adapted from the NHBS behavioral inventory and previously used with thousands of MSM by our team will collect information both on sexual behaviors with the main sex partner in the 3 months before the interview, and on sexual behaviors with all sex partners outside the relationship. For sex with the main partner, men will be asked to estimate the number of anal sex acts with the main partner, and the number of those acts that were condom-protected. For outside the relationship, we will ask a series of questions about each outside partner, including HIV status of that partner (if known), whether the sex outside the relationship was disclosed to the main partner, the number and type of sex acts with each outside partner, and the proportion of those sex acts that were protected by condoms.

SECONDARY OUTCOMES:
Linkage to Care | 6 months
  We will measure linkage to care with the following outcomes as indicators per the recent recommendations of the Institute of Medicine: within 3 months of HIV diagnosis (1) attending at least one clinical care appointment, (2) having at least one CD4 test performed, and (3) having at least one viral load test performed.

OTHER OUTCOMES:
Predisposing couple factors - Perceived Severity of HIV | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure predisposing couple factors one of which will be Perceived Severity of HIV scale. This construct involves the perception of the personal, psychosocial, and physical consequences of a particular health threat. We developed a total of 13 items that crossed three pertinent domains: personal, psychosocial and physical.
Predisposing couple factors - Preferences for General Lifestyle | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure predisposing couple factors. One factor of interest will be Preferences for General Lifestyle scale which includes 6 outcomes including diet and nutrition and social activities.
Predisposing couple factors - Preferences for General Sexual Health | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure predisposing couple factors. One factor of interest will be Preferences for Sexual Health Outcomes scale which relates to sexual health, for example, reducing your risk for HIV.
Predisposing couple factors - Conflict Style | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure predisposing couple factors. One factor of interest is Conflict Style which would determine how respondents typically handle conflict in their relationships using the Conflict Style Inventory.
Predisposing couple factors - Communication Style | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure predisposing couple factors. One factor of interest is Communication Style which would determine how respondents typically handle conflict in their relationships using the Conflict Style Inventory.
Predisposing couple factors - Problem-solving Skills | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure predisposing couple factors. One factor of interest is Problem-solving Skills which will be measured with the adherence problem solving / readiness scale.
Partner's transformation of motivation - Emotional Response | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure partner's transformation of motivation or the ability of the participants to respond (1) cognitively and (2) emotionally to the health threat. The scale for emotional response includes whether the respondent reports being fearful, nervous, or anxious about HIV.
Partner's transformation of motivation - Cognitive Response | 6 months
  Based on Lewis's model Couple's Interdependence Theory, we will measure partner's transformation of motivation or the ability of the participants to respond (1) cognitively and (2) emotionally to the health threat. The scale for cognitive response includes whether the respondent reports understanding the risks of HIV transmission associated with being in a sero-discordant relationship, and the risks associated with outside sex partners.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Stephenson, PhD, Principal Investigator — University of Michigan School of Nursing Department of Health Behavior and Biological Sciences
Locations (1):
- University of Michigan Center for Sexuality & Health Disparities (SexLab), Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stephenson R, Freeland R, Sullivan SP, Riley E, Johnson BA, Mitchell J, McFarland D, Sullivan PS. Home-Based HIV Testing and Counseling for Male Couples (Project Nexus): A Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 May 30;6(5):e101. doi: 10.2196/resprot.7341. PMID 28559225